CLINICAL TRIAL: NCT05974215
Title: Peri Implant Marginal Bone Height and Density Supporting Different Prosthesis Restoring Single Edentulous Mandible
Brief Title: Peri Implant Marginal Bone Height and Bone Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menatallah Mohamed Elhotieby (Other)
Responsible Party: Sponsor-Investigator, Menatallah Mohamed Elhotieby, researcher fixed and removable prosthodontics, National Research Centre, Egypt
Organization: National Research Centre, Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1431022023
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Implant Site Reaction
Keywords: Bone height; Bone density; Implant supported

STUDY DESIGN:
Intervention Model Description: group 1 mandibular implant supported overdenture group 2 mandibular implant supported fixed overdenture
Who Masked: Participant
Masking Description: each patient was not informed about type of received restoration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): patients received mandibular implant supported removable overdenture
  Interventions: Device: assessment of change in bone height by cone beam computed tomography
- group 2 (Active Comparator): patients received mandibular implant supported fixed overdenture
  Interventions: Device: assessment of change in bone height by cone beam computed tomography

INTERVENTIONS:
Device: assessment of change in bone height by cone beam computed tomography — bone height was measured at 1 ,30 ,90 days after denture insertion

SUMMARY:
This study aims to evaluate the effect of mandibular implant supported removable overdenture on bone height and density and compare it with implant supported fixed overdenture in single mandibular overdenture.

DETAILED DESCRIPTION:
In this study 10 patients will be selected following inclusion and exclusion criteria. In each group 5 patients (each patient will receive 6 implants) will be divided randomly into two groups.

Group I patients will receive mandibular implant supported removable overdenture, while Group II will receive mandibular implant supported fixed overdenture.

All patients will be given the usual home care instructions about wearing and caring of dentures and opposing arch. Regarding dentures, removal of them at night and cleaning with denture brush and mild soap will be required. Measurements of Bone height and Bone density will be obtained by using Cone Beam Computed Tomography (CBCT).

Measurements will be obtained at denture insertion, after 1 month and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker Patients
* Highly cooperative and motivated patients.
* Patients Systemically free from any immunosuppressive diseases.

Exclusion Criteria:

* Diabetic, hypertensive, cancer patients.
* Mandibular arch with thin knife edge, flat or flabby ridge, recent extractions and foreign bodies.
* Patients with temporo-mandibular joint disorders and bad oral habits.

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
assessment of change of bone height around dental implants | on the first day, on 30th day, 90th day
  bone height was assessed by cone beam computed tomography
assessment of change of bone density around dental implants | on the first day, on 30th day, 90th day
  bone density was assessed by cone beam computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Menatallah Elhotieby, Researcher, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Cairo, Egypt